CLINICAL TRIAL: NCT01301612
Title: A Phase II, Multicenter, Randomized,Two-Arm Clinical Study: An Investigational Arm Containing Nimotuzumab in Combination With Radiotion Therapy and Cisplatyn, and a Control Arm With Radiation Therapy and Cisplatin for the Definitive Treatment of Stage IB and IVA Uterine Cervical Carcinoma
Brief Title: Study of Nimotuzumab, Radiation Therapy and Cisplatin Versus Radiation Therapy and Cisplatin for Treatment of Stage IB e IVA UCC(CORUS)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Regulatory requirement. A phase III study is being designed.
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF 110
Record Dates: First submitted 2011-02-21; First posted 2011-02-23 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2012-01

CONDITIONS: Carcinoma; Adenocarcinoma; Uterine Cervix Adenosquamous Carcinoma
Keywords: carcinoma or adenocarcinoma or uterine cervix adenosquamous carcinoma
MeSH Terms: conditions — Carcinoma; Adenocarcinoma | interventions — nimotuzumab; Cisplatin; Brachytherapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiation therapy and Cisplatin (Active Comparator): Cisplatin, 40 mg/m2, IV - Weekly doses for 6 weeks Pelvic radiation therapy, 45 Gy External, Fractions of 1.8 Gy per day, 5 days a week Dose boosts,15 Gy ± 5%, External, Daily fractions of 1.8 Gy or 2 Gy per day, 5 days a week Brachytherapy (if indicaed), 40 Gy at spot A(low dose rate), Intracavitary 1 or 2 separate fractions for 1 to 3 weeks. 28 Gy at spot A, (high dose rate) Intracavitary,4 fractions of 7.0 Gy once or twice a week.
  Interventions: Drug: Cisplatin; Radiation: Radiation Therapy
- Nimotuzumab and (Experimental): Cisplatin, 40 mg/m2, IV, Weekly doses for 6 weeks.
  Nimotuzumab, 200 mg, Diluted into 250 mL of sodium chloride sterile solution 0.9% in intravenous infusion for 30 minutes, Weekly doses for 14 weeks.
  Pelvic radiation therapy, 45 Gy, External, Fractions of 1.8 Gy per day, 5 days a week.
  Dose boosts, 15 Gy ± 5%, External,Daily fractions of 1.8 Gy or 2 Gy per day, 5 days a week
  Brachytherapy (In case there is indication, should it be performed, not to be longer than the expected 70 days for the entire radiation therapy), 40 Gy at spot A (low dose rate) Intracavitary 1 or 2 separate fractions for 1 to 3 weeks 28 Gy at spot A (high dose rate), Intracavitary, 4 fractions of 7.0 Gy once or twice a week.
  Interventions: Drug: Nimotuzumab; Drug: Cisplatin; Radiation: Brachytherapy

INTERVENTIONS:
Drug: Nimotuzumab — Nimotuzumab, 200 mg, IV, Weekly doses for 14 weeks
  Arms: Nimotuzumab and
Drug: Cisplatin — Cisplatin, 40 mg/m2, IV, Weekly doses for 6 weeks
  Arms: Nimotuzumab and
Radiation: Brachytherapy — Brachytherapy: 40 Gy at spot A(low dose rate, Intracavitary, 1 or 2 separate fractions for 1 to 3 weeks.
  Brachytherapy: 28 Gy at spot A (high dose rate), Intracavitary 4 fractions of 7.0 Gy once or twice a week.
  Arms: Nimotuzumab and
Drug: Cisplatin — Cisplatin, 40 mg/m2, IV. Weekly doses for 6 weeks
  Arms: Radiation therapy and Cisplatin
Radiation: Radiation Therapy — Pelvic radiation therapy: 45 Gy, External, Fractions of 1.8 Gy per day, 5 days a week.
  Dose boosts: 15 Gy ± 5%, External, Daily fractions of 1.8 Gy or 2 Gy per day, 5 days a week.
  Brachytherapy 40 Gy at spot A(low dose rate.) Intracavitary 1 or 2 separate fractions for 1 to 3 weeks.
  28 Gy at spot A (high dose rate, Intracavitary, 4 fractions of 7.0 Gy once or twice a week
  Arms: Radiation therapy and Cisplatin

SUMMARY:
The primary study objective will be to assess the efficacy of the combination of radiation therapy with nimotuzumab and cisplatin, as compared to the combination of radiation therapy plus cisplatin in the treatment of Uterine Cervical Carcinoma (UCC).

The secondary study objectives will be safety and tolerability evaluations, to determine treatment feasibility and the interim efficacy evaluation according to other parameters routinely used in oncology.

DETAILED DESCRIPTION:
This will be a phase II, randomized, controlled, open-label, multicenter, and two-arm study. The study will be conducted in Brazil and has the purpose of determining the activity and safety of nimotuzumab in terms of overall and distant disease-free survival, radiological and clinical gynecological examinations, as well as by biopsy, if indicated, progression-free survival, local control of long-term disease, frequency of treatment-emergent adverse events, frequency of severe treatment-emergent adverse events.

All participating patients will sign a consent form before they undergo any study-related procedure.The eligible patients will have stage IB and IVA uterine cervical carcinoma and they will be randomized to one of two treatment groups.

Randomization and treatment assignment will be performed by a company specifically contracted for such purpose and will be per research site and disease stage (IB2 to IIIA versus IIIB to IVA), 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Diagnosis of histologically confirmed stages IB2 (> 4 cm) to IVA prickle-cell carcinoma or adenocarcinoma or uterine cervix adenosquamous carcinoma, according to FIGO system,7 (see Appendix A for guidance about staging);
* Measurable disease according to RECIST 1.139 or at least disease evaluable through imaging methods and/or gynecological examination (magnetic resonance imaging (MRI) scans within six weeks prior to randomization will be accepted, computed tomography will accepted in case MRI is contraindicated);
* Indication of definitive treatment with chemotherapy and radiation therapy, at the investigator's discretion;
* Performance status < 2, according to the Eastern Cooperative Oncology Group criteria 40 (ECOG; see Appendix C);
* Adequate body functions, indicated by:Serum creatinine < 1.2 mg/100 mL; Creatinine clearance > 60 mL/min (estimate); Bilirubin up to 1.5-fold the upper limit of normal (ULN) and transaminases, alkaline phosphatase and gamma-glutamyltransferase up to 2.5-fold the ULN; Leucocytes > 3,000/μL; Neutrophils > 1,500/μL; Hemoglobin > 10 g/dL; Platelets > 80,000/μL;
* Signed informed consent form.

Exclusion Criteria:

* Para-aortic lymph nodes involvement through radiological and/or surgical staging, at investigator's discretion;
* Current severe comorbidity that, in the investigator's opinion, would put the patient at a significantly higher risk or will jeopardize protocol compliance;
* Current bowel inflammatory disease;
* Current major neurological or psychiatric disease, including clinically significant dementia and seizures, at the investigator's discretion;
* Known hypersensitivity or allergic reactions to study treatment;
* Current uncontrolled hypercalcemia (> 11,5 mg/dL, that is, grade > 1 according to Common Terminology Criteria for Adverse Events [CTCAE] v4.02, of US National Cancer Institute)41;
* Know HIV positive status (enrollment of patients with hepatitis B or C is at the investigator's discretion);
* Pregnancy or lactation;
* Female patients, as well as their partners, who wish to become pregnant or are unwilling to use an appropriate contraceptive method throughout the study period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Local control of disease | 1 year
  Local control of disease will be measured by magnetic resonance imaging (MRI), clinical gynecological examinations, as well as by biopsy (if indicated), 12 weeks after treatment end.

SECONDARY OUTCOMES:
Complete clinical response rate | 3 years
  * Overall survival;
  * Distant disease-free survival;
  * Progression-free survival;
  * Local control of long-term disease; Frequency of treatment-emergent adverse events; o Frequency of severe treatment-emergent adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Lago, Principal Investigator — Núcleo de Novos Tratamentos em Câncer - NNTC
Locations (7):
- Brazil (7):
  - Centro de Pesquisa Clínica da Liga Norte Riograndense contra o Câncer, Natal, Rio Grande do Norte
  - Hospital de Caridade de Ijui - ONCOSITE Centro de Pesquisa Clínica em Oncologia, Ijuí, Rio Grande do Sul
  - Hospital Santa Rita - Núcleo de Novos Tratamentos em Câncer, Porto Alegre, Rio Grande do Sul
  - Caism - Unicamp, Campinas, São Paulo
  - Centro de Pesquisas Clínicas da Fundação Amaral Carvalho, Jaú, São Paulo
  - ICESP, São Paulo, São Paulo
  - Hospital Santa Marcelina, São Paulo, São Paulo